CLINICAL TRIAL: NCT05455437
Title: Monitoring and Evaluation Study of Project ECHO for ILD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Pulmonary Care and Research Collaborative Limited (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ILDC-002
Record Dates: First submitted 2022-06-30; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Interstitial Lung Diseases
Keywords: Progressive Fibrosing Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis; Interstitial Lung Disease Associated With Systemic Sclerosis; Myositis-Associated Interstitial Lung Disease; Sarcoidosis; Hypersensitivity Pneumonitis; Pulmonary Fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis; Sarcoidosis; Alveolitis, Extrinsic Allergic; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will utilize pre-post survey measures to evaluate Project ECHO for ILD with respect to an initial set of practice and clinical outcomes and relies on questionnaire data obtained from providers participating in Project ECHO for ILD at baseline, at 6 months, and at study end.

DETAILED DESCRIPTION:
Project ECHO (Extension for Community Healthcare Outcomes) is a knowledge-sharing model to expand the capacity of the health care workforce so that more people can get high quality care for their health conditions in or near the communities where they live. The model brings specialty disease expertise to community providers through its hub-and-spoke networks. The model relies on videoconferencing to connect local providers in non-urban or underserved communities (spoke sites) with an interdisciplinary team of specialist providers at academic medical centers (hubs) during virtual "teleECHO" clinic sessions, which include brief educational lectures and case-based, experiential learning. It is a guided, technology-enabled collaborative practice model in which community providers become experts in an area of community need within the scope of their practice, operating with increasing independence as their skills and self-efficacy grow. The model establishes meaningful, ongoing relationships with hub specialists who serve as telementors for spoke providers and relies on case-based learning from presentations of real-world de-identified patient cases.

The overarching goal of the project is to implement and evaluate an adaptation of the ECHO model to interstitial lung disease (ILD) diagnosis and care among primary care physicians (PCPs) and community pulmonologists in non-urban or underserved communities.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonologists and primary care physicians who participate in Project ECHO for ILD.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pulmonologists and primary care physicians who participate in Project ECHO for ILD.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Impact on procedural knowledge | Up to 18 months
  Change in participants' skills or competence in knowing ILD testing and treatment procedures based on a Likert scale rating (1=no skill and 7=expert, teach other) included in the structured participant surveys administered at baseline, 6 months, and at study end.
Impact on local care utilization | Up to 18 months
  Change of proportion of patients utilizing local ILD care services, including the frequency of local follow-up visits and testing. Change in scores will be calculated between structured participant surveys responses at baseline, 6 months, and at study end.

SECONDARY OUTCOMES:
Time to ILD diagnosis | Up to 18 months
  The amount of time it takes for a participant's patient to be given an established, named ILD diagnosis (IPAF, IPF, HP, CTD-ILD, myositis-ILD, idiopathic NSIP, etc.) from onset of respiratory symptoms and from the time of first pulmonologist appointment. This data will be obtained from teleECHO clinic management records and participants' case and follow-up reporting for patients who were presented to the ECHO for diagnosis.
Content expert facilitation | Up to 18 months
  Proportion of participants who agree that the quality of content expert facilitation was adequate during the teleECHO session. This will be collected monthly from post-session surveys via a Likert scale (1=strongly disagree and 5=strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa Barakat, PhD, Principal Investigator — Pulmonary Care and Research Collaborative, Ltd.
Locations (1):
- Pulmonary Care and Research Collaborative, Ltd., Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No